CLINICAL TRIAL: NCT05677256
Title: A Phase IV Open-label, Randomized, Parallel-group Study to Evaluate Pharyngeal Immunity to Poliovirus Type-2 in Healthy bOPV- Versus IPV-vaccinated Infants
Brief Title: A Study to Evaluate Pharyngeal Immunity to Poliovirus Type-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPV-005-ABMG
Record Dates: First submitted 2022-12-09; First posted 2023-01-10 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPV-primed Group (Experimental): Approximately 250 subjects to receive 3 doses of IPV administered at approx. 6, 10, 14 weeks of age and an nOPV2-002 challenge at approx. 18 weeks of age.
  Interventions: Biological: nOPV2
- bOPV-primed Group (Active Comparator): Approximately 250 subjects to receive 3 doses of bOPV administered at approx. 6, 10, 14 weeks of age and an nOPV2-002 challenge at approx. 18 weeks of age.
  Interventions: Biological: nOPV2

INTERVENTIONS:
Biological: nOPV2 — Vaccination

SUMMARY:
The study will compare the poliovirus type-2 pharyngeal mucosal excretion in the first week, and at 2 and 4 weeks following the administration of a challenge novel OPV2 (nOPV2) dose at 18 weeks of age in 2 parallel groups of infants

DETAILED DESCRIPTION:
In the light of the switch from OPV to IPV and the continued presence of cVDPV2 in many countries, it is important to understand and quantify the impact of IPV on pharyngeal mucosal immunity, to inform whether and to what extent the mucosal and humoral immune response following IPV could reduce transmission and spread.

This study will assess the effect of vaccination with IPV in parallel with poliovirus type-2 naïve infants (infants having received bOPV) on the pharyngeal and fecal shedding and the induction of immunity following type-2 poliovirus challenge. This understanding would provide critical information on the potential use of IPV in specific settings to interrupt transmission / reduce spread. The results from this study may potentially have important consequences on public health policy in countries which use IPV for infant priming, as they will help to show the extent to which a type-2 mucosal immunity gap remains following a primary series of IPV.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 6 to 8 weeks with birth weight >2,500 g.
2. Healthy infants without obvious medical conditions like immunodeficiency diseases, severe congenital malformations, severe neurological diseases or any other disease that require high doses of corticosteroids or immunotherapies that preclude the subject from participating in the study as established by the medical history and physical examination.
3. Written informed consent obtained from both parents or legal guardian(s) as per country regulations.

Exclusion Criteria:

1. Infants who have received previous vaccination against poliomyelitis.
2. Any confirmed or suspected immunosuppressive or known immunodeficient condition including human immunodeficiency virus infection in the potential participant or any member of the subject's household.
3. Family history of congenital or hereditary immunodeficiency.
4. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
5. Known allergy to any component of the study vaccines or to any antibiotics that share molecular composition with a component of the study vaccines.
6. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections (of IPV)
7. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
8. Acute severe febrile illness on the day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all inclusion criteria are met.).
9. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.
10. Infants from multiple births or born prematurely (< 37 weeks of gestation).

Ages: 5 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Poliovirus type-2 viral shedding | 1 month
  To compare the presence of poliovirus type-2 in pharyngeal samples detected by reverse-transcription polymerase chain reaction (RT PCR) in the first week, and at D14 and D28 in both groups.

SECONDARY OUTCOMES:
Pharyngeal neutralizing antibodies (NAbs) and IgA response to poliovirus type-2. | 1 month
  To assess and compare the pharyngeal NAbs activity, and poliovirus type-2-specific concentrations of pharyngeal mucosal immunoglobulin A (IgA) on D0, D14 and D28 in both groups.
Seroconversion rate of poliovirus type-2 neutralizing antibodies (NAbs) | 2 months
  To assess the cummulative seroconversion (SC) rate of poliovirus type-2 NAbs on D28 and D56 following administration of a challenge dose of nOPV2 in both groups.Seroconversion is defined as seropositive (titer ≥1:8) in those initially seronegative, or among those initially seropositive, as a minimum 4-fold higher titer (and seropositivity) than that which is expected due to maternal antibodies.
Incidence of Serious Adverse Events (SAEs) and Important Medical Events (IMEs) | 5 months
  To assess the number of subjects experiencing SAEs and IMEs following administration of IPV, bOPV and nOPV2 throughout the whole study period.

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Diseases Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No